CLINICAL TRIAL: NCT03094741
Title: Evaluation of a Mobile Digital Solution for Cancer Care and Research: A Feasibility Study
Brief Title: Evaluation of a Mobile Digital Solution for Cancer Care and Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: CancerLife (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: JWCI-17-0301
Record Dates: First submitted 2017-03-21; First posted 2017-03-29 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cancer; Caregivers; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CancerLife Feasibility Group (Experimental): Participants will be recruited through advertisements targeted to a specific audience using the keywords cancer and cancer survivors
  Interventions: Other: CancerLife

INTERVENTIONS:
Other: CancerLife — CancerLife is a mobile digital solution that allows patients to broadcast their health status inside a private invitation only group, text, email or publicly in Facebook or Instagram. By doing, so the patient collects his/her own patient-reported outcomes data and then share this data with their doctor or care team.

SUMMARY:
The primary purpose of this pilot study is to evaluate the feasibility and acceptability of a Mobile Digital Solution in monitoring and collecting symptom burden data. The proposed study is meant to be the preparatory work for an intervention study to test the effect of Mobile Digital Solutions on improving patient outcomes by prompting early interventions for symptom relief and support of patient and family caregiver quality of life (QOL).

DETAILED DESCRIPTION:
Demographic information and patient-reported symptoms will be collected from study participants through a mobile health application called CancerLife that they can download (FREE) from their mobile device app store (Android or iOS). Participants will be asked to broadcast their emotional and physical status through a list of symptom list within the app as well as how that symptom is impacting their quality of life and activities of daily living. This data will be collected inside the application and display in easy to understand pie charts. Participants will also have the option to broadcast their entry to their social network.

Since the objective of the current feasibility study is to evaluate the feasibility and acceptability of a Mobile Digital Solution in monitoring and collecting symptom burden and QOL data, the investigators will include a standard validated instrument (FACT-G: Functional Assessment of Cancer Therapy - General) as part of this study. Participants will be asked to complete the FACT-G after initial registration and weekly for up to 4 weeks. Participants will receive electronic mail messages with a link to CancerLife weekly as a reminder to access the website.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of cancer
* Karnofsky Index ≥50%
* Age > 18 years

Exclusion Criteria:

* Relevant cognitive impairment
* Insufficient knowledge of English language to complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Feasibility/ Participation Rate | 4 weeks
  number of individuals who participate in the study divided by the number of individuals who opened the link

SECONDARY OUTCOMES:
Open Rate | 4 weeks
  number of individuals who open the link divided by total number of individuals reached by the advertisement
Refusal rate | 4 weeks
  number of individuals who declined to participate divided by the number of individuals who opened the link
Retention rate | 4 weeks
  number of mission data divided by total number of items available
Rate of missing data | 4 weeks
  number of mission data divided by total number of items available
Participant Satisfaction | 4 weeks
  describe the usability, satisfaction, and desirability of the Mobile Digital Solution using a patient experience survey at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Study Chair — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No